CLINICAL TRIAL: NCT01573949
Title: A Pilot Study: Metformin Therapy in Heart Failure Patients With Early Diabetes or at High Risk of Developing Diabetes (Pre-Diabetes)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tamara Horwich, Tamara Horwich, MD, MS, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-002909
Record Dates: First submitted 2012-03-29; First posted 2012-04-10 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Diabetes; Heart Failure
Keywords: Heart Failure; Diabetes; Pre-diabetes; Early type II diabetes; Metformin; Pharmacotherapy with metformin for prevention of DM in HF patients with pre-diabetes (pre-DM) and glycemic control in HF patients with early type II DM
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Metformin will be started at 500 mg PO BID and pending lab values may be titrated to 1000 mg PO BID at 1 month.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be started at 500 mg PO BID and pending lab values may be titrated to 1000 mg PO BID at 1 month for a duration of 3 months.

SUMMARY:
The Ahmanson-UCLA Cardiomyopathy Center is conducting a clinical research study that will assess the use of the medication metformin to improve quality of life, exercise capacity, and improved outcomes in heart failure patients with pre-DM or early DM (type II).

If the patient participates in this study, the patient will receive the drug metformin for approximately 3 months. During the study the patient will undergo comprehensive testing which includes blood draws and echocardiograms. The patient will also fill out a questionnaire. The patient must be 18 years old to participate.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic HF of any etiology
* age ≥ 18 years
* fasting blood sugar equal or greater than 100 mg/dL, or pre-DM (HbA1c 5.7 - 6.4%) or early DM (HbA1c ≥ 6.5%)

Exclusion Criteria:

* current metformin therapy or other anti-diabetic therapy
* previous intolerance to metformin therapy
* renal dysfunction (Cr >1.5 in men or > 1.4 in women or creatinine clearance < 60 ml/minute)
* history of lactic acidosis
* current or planned pregnancy or breast-feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Horwich, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ahmanson-UCLA Cardiomyopathy Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin at 500 mg PO BID and pending lab values may have been titrated to 1000 mg PO BID at 1 month.
Period: Overall Study
Arm/Group | Metformin
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Health-Related Quality of Life (HRQoL)
Description: HRQoL as assessed by the Minnesota Living With Heart Failure Questionnaire (MLHFQ)
  The MLHFQ is a self-administered questionnaire for patients with HF, comprising 21 items rated on six-point Likert scales, representing different degrees of impact of HF on HRQoL, from 0 (none) to 5 (very much). It provides a total score range 0-105. Lower scores indicate better health-related quality of life (HRQoL).
Time Frame: 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Metformin
Number analyzed (Participants) | 7
score on a scale
  Baseline | 37 [1 to 91]
  Three Months | 37 [6 to 86]

2. Secondary Outcome: Glycated Hemoglobin (HbA1c)
Description: The HbA1c test measures how much glucose is bound to hemoglobin in the red blood cells. The test shows the average level of glucose in blood for the past 3 months (the average lifespan of red blood cells). If glucose levels have been high over recent weeks, the hemoglobin A1c test will be higher.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Metformin
Number analyzed (Participants) | 7
percentage of glycated hemoglobin
  Baseline | 6.1 (0.4)
  Three Months | 6.2 (0.4)

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Obtained from Echocardiography
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Metformin
Number analyzed (Participants) | 7
percent ejection fraction
  Baseline | 25 (8)
  Three Months | 26 (9)

4. Secondary Outcome: Creatinine Level as a Measure of Renal Function
Description: Serum creatinine
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin
Number analyzed (Participants) | 7
mg/dL
  Baseline | 1.1 (0.2)
  Three Months | 1.1 (0.2)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes